CLINICAL TRIAL: NCT06577701
Title: Respiratory Disease Cohort Studies of Chinese Medicine for Chronic Obstructive Pulmoriary Disease (RESEARCH-COPD)
Brief Title: Respiratory Disease Cohort Studies of Chinese Medicine for COPD(RESEARCH-COPD)
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RESEARCH-COPD
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmoriary Disease (COPD); Preserved Ratio Impaired Spirometry (PRISM)
Keywords: Chronic Obstructive Pulmoriary Disease (COPD); Preserved Ratio Impaired Spirometry (PRISM); Complication (medicine); Traditional Chinese Medicine; Registration; Cohort study
MeSH Terms: interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Traditional Chinese Medicine cohort: Regulated use of Chinese medicine treatment protocols is included as an exposure factor. Continuous medication for more than 3 months per year, or intermittent medication for more than 6 months per year was the exposure group (TCM diagnosis and treatment plan cohort).
  Interventions: Drug: traditional Chinese medicine (TCM)
- Non Traditional Chinese Medicine cohort: Other patients who did not fit into the TCM group.
  Interventions: Drug: non traditional Chinese medicine (non-TCM)

INTERVENTIONS:
Drug: traditional Chinese medicine (TCM) — Regulated use of Chinese medicine treatment protocols is included as an exposure factor. Exposure was defined as taking the medication continuously for more than 3 months per year, or taking the medication intermittently for more than 6 months per year. According to the standardised use of TCM protocols, the group was divided into an exposed group (TCM protocols cohort) and a non-exposed group (non-TCM protocols cohort).
  Groups: Traditional Chinese Medicine cohort
Drug: non traditional Chinese medicine (non-TCM) — Regulated use of Chinese medicine treatment protocols is included as an exposure factor. Exposure was defined as taking the medication continuously for more than 3 months per year, or taking the medication intermittently for more than 6 months per year. According to the standardised use of TCM protocols, the group was divided into an exposed group (TCM protocols cohort) and a non-exposed group (non-TCM protocols cohort).
  Groups: Non Traditional Chinese Medicine cohort

SUMMARY:
This study will establish a registration research platform, a clinical research database and a biospecimen bank for the prevention and treatment of COPD with Chinese medicine. Based on the COPD registry database, a cohort of Chinese medicine for COPD prevention and treatment will be established.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common chronic respiratory disease with high prevalence, high mortality rate, high disability rate and heavy disease burden, seriously endangering people's health. The prevalence of COPD among people aged 40 and above in China is 13.7%, with nearly 100 million patients. The situation of high prevalence, high mortality, and high disability is not matched by the low awareness rate, low lung function test rate, and low treatment rate, which is a serious situation for prevention and control. 2021 edition of 'Global Initiative on Chronic Obstructive Lung Disease (GOLD)' puts forward the concept of pre-COPD, which indicates that the concept of prevention and treatment of COPD has begun to change to prevention and early intervention, and is also related to the concept of intermediate medicine. The concept of pre-COPD has been proposed in the 2021 edition of GOLD, indicating that the concept of prevention and treatment of COPD has begun to shift towards prevention and early intervention, which is also in line with the idea of 'treating the disease before it is diagnosed' in TCM. Chinese medicine has certain advantages in the prevention and treatment of COPD. Currently, there is a lack of TCM diagnostic and treatment protocols for the early stage of COPD, and TCM diagnostic and treatment protocols for the stable stage of COPD need to be optimised. Therefore, based on the Chinese COPD registry management system, this study took the pre-CPD population and stable stage patients as the research object, and used the standardised use of Chinese medicine diagnostic and treatment protocols as the exposure factor to carry out a multicentre prospective cohort study, with a follow-up of 2 years, using the morbidity rate, the rate of decline in lung function FEV1, etc., to evaluate the efficacy of Chinese medicine diagnostic and treatment protocols for pre-COPD, and using the rate of occurrence of acute exacerbation, The efficacy of TCM treatment protocols for patients with stable COPD was further evaluated using the incidence of acute exacerbation and quality of survival. This will provide high-quality evidence-based medical evidence for the prevention and treatment of COPD by TCM.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for chronic obstructive pulmonary disease (COPD) or preserved ratio impaired spirometry (PRISm).
* Age ranges from 18 years to 80 years.
* The investigators agreed to participate in this clinical study by voluntarily signing an informed consent form.

Exclusion Criteria:

* Patients with delirium, dementia, various mental illnesses.
* Pregnant and planned pregnant or lactating women.
* Patients with other serious systemic diseases.
* Patients who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease (COPD) is a major disease that poses a serious threat to public health, with a prevalence rate of 13.7% in China for people aged 40 years and older, and a prevalence rate of 20.51% in high-risk groups, with a prevalence rate of COPD in high-risk groups of 33.39%, Early screening and identification are of great significance in delaying the progression of lung function and reducing the incidence of COPD. At the same time, patients with COPD are often comorbid with other diseases, and comorbidities have a significant impact on disease progression, consultation, hospitalization, morbidity and mortality, requiring more standardized and systematic recommendations to guide clinical practice.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Frequencies of acute exacerbations (AEs) | Frequency of acute exacerbations at months 3, 6, 9, 12, 15, 18, 21, and 24.
  The frequencies of acute exacerbations (AEs) will be recorded.
Incidence of COPD | 24 months after enrollment.
  The incidence of COPD will be recorded.

SECONDARY OUTCOMES:
6 Six Minute Walk Distance (6MWD) | 6MWD at months 3, 6, 9, 12, 15, 18, 21, and 24.
  6MWD will be applied to evaluate the exercise capacity. The higher values indicate the better exercise capacity.
Traditional Chinese medicine syndromes | The Traditional Chinese medicine syndromes at months 3, 6, 9, 12, 15, 18, 21, and 24.
  The Traditional Chinese medicine syndromes will be recorded.
Forced expiratory volume in one second (FEV1) | Change from baseline FEV1 at months 6, 12, 18 and 24.
  FEV1 will be applied to assess pulmonary function.
Forced vital capacity (FVC) | Change from baseline FVC at months 6, 12, 18 and 24.
  FVC will be applied to assess pulmonary function.
FVC as the percentage of the predicted value (FVC%) | Change from baseline FVC% at months 6, 12, 18 and 24.
  FVC% will be applied to assess pulmonary function.
Forced expiratory volume in one second / forced vital capacity (FEV1/FVC) | Change from baseline FEV1/FVC at months 6, 12, 18 and 24.
  FEV1/FVC will be applied to assess pulmonary function.
Diffusing capacity of the lungs for carbon monoxide (DLCO) | Change from baseline DLCO at months 6, 12, 18 and 24.
  DLCO will be applied to assess pulmonary function.
COPD Assessment Test (CAT) | At months 6, 12, 18 and 24.
  CAT will be applied to assess quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China